CLINICAL TRIAL: NCT00917514
Title: An Investigational Study to Test Usability of the Electronic Dosing Equipment Medicpen During Azathioprine Treatment in Patients With Crohn's Disease or Ulcerative Colitis
Brief Title: An Investigational Study to Test Usability of the Electronic Dosing Equipment Medicpen
Status: Completed | Type: Observational
Sponsor: Medicpen AB (Industry)
Responsible Party: CEO Cristian Hallin, MedicPen AB
Other Study IDs: MP-01
Record Dates: First submitted 2009-06-09; First posted 2009-06-10 (Estimated); Last update posted 2010-02-26 (Estimated); Status verified 2009-06

CONDITIONS: Crohn's Disease; Ulcerative Colitis
Keywords: Dosing Tool; Compliance; User Friendly; Crohn's Disease; Ulcerative Colitis
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Patient Compliance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a study of the electronical dosing tool MedicPen and it's qualities with regards to user friendliness and medication compliance.

DETAILED DESCRIPTION:
The medical device MedicPen will be investigated for it's qualities with regards to medication compliance and user friendliness. The patient group selected here is patients with Crohn's disease that are treated with Azathioprine. The patient selection was made since the metabolite can be easily measured and the compliance can be therefore be followed. The treatment will follow the standard care given to these patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 18 years or older
* Provided written informed consent
* Diagnosed with Chron's disease or Ulcerative Colitis
* Treated with Azathiprine for at least 6 months prior to study start

Exclusion Criteria:

* Patients who are, for some reason, judged by the responsible investigator to be unable to handle the device to be tested.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Chrohn's disease or Ulcerative Colitis. Male or Female above 18 years of age. Ability to provide written informed consent. Must have been on Azathioprine treatment for at least 6 months prior to study start.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2009-06; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
User friendliness of Dosing Tool MedicPen | June 2009 to Nov 2009

SECONDARY OUTCOMES:
Measure treatment compliance | June 2009 to Nov 2009

CONTACTS AND LOCATIONS:
Overall Officials: Mikael Lördal, Cheif MD, Principal Investigator — Department for Gastrointestinal Medicine, Karolinska University Hospital, Huddinge
Locations (1):
- Department for Gastrointestinal medicin Karolinska University Hospital, Huddinge, Sweden